CLINICAL TRIAL: NCT02468063
Title: A Prospective Study to Assess the Efficacy of Early Introduction of a Combination of Low Dose Vasopressin Analogue in Addition to Noradrenaline as a Vasopressor in Patients of Cirrhosis With Septic Shock
Brief Title: To Assess the Efficacy of Early Introduction of a Combination of Low Dose Vasopressin Analogue in Addition to Noradrenaline as a Vasopressor in Patients of Cirrhosis With Septic Shock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-001
Record Dates: First submitted 2015-05-22; First posted 2015-06-10 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-01

CONDITIONS: Cirrhosis With Septic Shock
MeSH Terms: interventions — Terlipressin; Norepinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Noradrenaline + low dose terlipressin (Experimental)
  Interventions: Drug: Low dose terlipressin; Drug: Noradrenaline
- Noradrenaline (Active Comparator)
  Interventions: Drug: Noradrenaline

INTERVENTIONS:
Drug: Low dose terlipressin — Terlipressin-2mg (low dose )
  Arms: Noradrenaline + low dose terlipressin
Drug: Noradrenaline — Noradrenaline at 7.5 mcg/min, maximum of 60mcg/min. stepped up every 15 min
  Arms: Noradrenaline + low dose terlipressin
Drug: Noradrenaline — Noradrenaline- 3.75 mcg/min to 30 mcg/min. stepped up every 15 min
  Arms: Noradrenaline

SUMMARY:
The consecutive patients admitted to Intensive care unit of Hepatology department of ILBS and full filling all the eligibility criteria will be enrolled in 1:1 ration by the process of randomization.- The study is an open level study. The investigators will strictly follow the randomization table to give therapy as per the intervention arm.

* Intervention:-the therapeutic intervention is vasopressor i.e. noradrenaline alone and terlipressin along with noradrenaline to maintain the MAP >65mm Hg.
* Intervention arm

  * Arm (A) - Noradrenaline
  * Arm (B) - Noradrenaline + low dose terlipressin

ELIGIBILITY:
Inclusion Criteria:

* 18-70 yr
* Cirrhosis with septic shock not responding to fluid resuscitation within 2 hrs.

Exclusion Criteria:

* ECG (ElectroCardiography)changes at presentation which exclude the use of vasopressin analouges
* Cardiac dysfunction ( valvular heart disease, coronary artery disease)
* Acute mesenteric ischemia (confirmed or suspected) or vasospastic diathesis (e.g. Reynaud's syndrome or related diseases).
* Pregnancy
* Acute GI bleed
* No Consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Target MAP (Mean Arterial Pressure) >65 mm Hg at 6 hrs | 6 hours

SECONDARY OUTCOMES:
Maintenance of target MAP (Mean Arterial Pressure) | 2 days
  MAP is Mean Arterial pressure SVR is Sustained Virologic Response
Survival | 28 days
Survival | 48 hours
Microcirculation (lactate level, Lactate clearance, SCVO2, ABG-VBG Pco2 difference), | 2 years
Tissue perfusion (lactate level, Lactate clearance, SCVO2, ABG-VBG Pco2 difference), | 2 years
Effect on - AKI (Acute kidney Injury), | 2 years
Effect on variceal bleed | 2 years
Effect on rebound hypotension | 2 years
Effect on organ failure | 2 years
Length of ICU | 2 years
Length of hospital stay. | 2 years
Incidence of adverse events. | 2 years
Predictors of adverse events. | 2 years
SVR (Sustained Virologic Response) ≥600 at 48 hrs | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Vikash Prakash, MD, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India